CLINICAL TRIAL: NCT02998684
Title: Learning Enhancement Through Neurostimulation in Autism
Acronym: LENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00056912
Record Dates: First submitted 2016-12-01; First posted 2016-12-20 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Autism
Keywords: Autism; Adolescent; Social skills
MeSH Terms: conditions — Autistic Disorder; Social Skills

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Transcranial Direct Current Stimulation (Active Comparator): Participants will receive active Transcranial Direct Current Stimulation
  Interventions: Device: Active Transcranial Direct Current Stimulation; Behavioral: PEERS Social Skills Training
- Sham Transcranial Direct Current Stimulation (Sham Comparator): Participants will receive sham Transcranial Direct Current Stimulation
  Interventions: Device: Sham Transcranial Direct Current Stimulation; Behavioral: PEERS Social Skills Training

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation
  Arms: Active Transcranial Direct Current Stimulation
Device: Sham Transcranial Direct Current Stimulation
  Arms: Sham Transcranial Direct Current Stimulation
Behavioral: PEERS Social Skills Training — 14 weekly social skills training sessions for all participants

SUMMARY:
This study will examine whether brain stimulation paired with social skills learning can help teenage boys with autism learn how to make and keep friends. Brain stimulation can enhance learning in some people. This study involves enrolling in a 14-week training program where teenage boys with autism interact in small groups and learn social skills. During the 14-week program participants will receive active brain stimulation, or non-active stimulation (placebo). Before and after this training, MRI scans will be taken to see whether the training with active brain stimulation made a different in brain activation.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder

Exclusion Criteria:

* Intellectual Disabilities (Full-scale IQ <70)
* Hx of seizures within the last one year
* Contraindications for fMRI, such as metal implants in the head

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Joseph, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical Univeristy of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Transcranial Direct Current Stimulation: Participants will receive active Transcranial Direct Current Stimulation
  Active Transcranial Direct Current Stimulation
  PEERS Social Skills Training: 14 weekly social skills training sessions for all participants
- Sham Transcranial Direct Current Stimulation: Participants will receive sham Transcranial Direct Current Stimulation
  Sham Transcranial Direct Current Stimulation
  PEERS Social Skills Training: 14 weekly social skills training sessions for all participants
Period: Overall Study
Arm/Group | Active Transcranial Direct Current Stimulation | Sham Transcranial Direct Current Stimulation
Started | 7 | 7
Completed | 4 | 6
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Transcranial Direct Current Stimulation | Sham Transcranial Direct Current Stimulation | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 13
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 5 | 10
  Black/African American | 0 | 2 | 2
  Hispanic | 1 | 0 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Test of Adolescent Social Skills Knowledge (TASSK)
Description: Change in TASSK raw scores from pre- to post-treatment, i.e., baseline to 14-weeks (Post minus pre-treatment: positive scores indicate improvement). Assessment scores can range from 0 to 26, 0 being the lowest possible score and 26 being the highest.
Time Frame: Baseline to 14-weeks
Population: Number of participants who completed study questionnaire pre and post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcranial Direct Current Stimulation | Sham Transcranial Direct Current Stimulation
Number analyzed (Participants) | 3 | 6
score on a scale | 8 (2) | 3.5 (2.1)

2. Primary Outcome: Social Responsiveness Scale (SRS)
Description: Change in SRS raw scores from pre- to post-treatment, i.e., baseline to 14-weeks (Pre minus post-treatment: positive scores indicate improvement). Raw scores range from 0 to 195, with higher scores indicating greater severity of symptoms.
Time Frame: Baseline to 14 weeks
Population: Data for participants who completed all 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcranial Direct Current Stimulation | Sham Transcranial Direct Current Stimulation
Number analyzed (Participants) | 4 | 6
score on a scale | 23.5 (18.2) | 26.5 (22.6)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Active Transcranial Direct Current Stimulation | Sham Transcranial Direct Current Stimulation
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT02998684/Prot_SAP_000.pdf